CLINICAL TRIAL: NCT00426933
Title: Phase 2 Multicenter Randomized Semi-Single Blind Study to Compare Efficacy and Safety of High-dose Short Duration Daptomycin With Conventional Therapy in Complicated Skin and Skin Structure Infections Due to Gram-positive Bacteria
Brief Title: Phase 2 Safety and Efficacy Study of Daptomycin in Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: A. Wheeler, Cubist Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAP-HDSD-06-01
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Soft Tissue Infections
Keywords: cSSSI; MRSA
MeSH Terms: conditions — Soft Tissue Infections | interventions — Daptomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daptomycin
Drug: Vancomycin

SUMMARY:
multicenter, randomized (1:1), semi-single blind study comparing the safety and efficacy of HDSD daptomycin (10 mg/kg q24h for 4 days) with that of comparator (vancomycin +/- SSP for 7-14 days) in patients with cSSSI due to Gram-positive bacteria. Patients will be randomized on a 1:1 basis to receive either daptomycin 10 mg/kg i.v. q24h for 4 days or vancomycin 1 g. q12h for up to 14 days.

DETAILED DESCRIPTION:
multicenter, randomized (1:1), semi-single blind study comparing the safety and efficacy of HDSD daptomycin (10 mg/kg q24h for 4 days) with that of comparator (vancomycin +/- SSP for 7-14 days) in patients with cSSSI due to Gram-positive bacteria. Patients will be randomized on a 1:1 basis to receive either daptomycin 10 mg/kg i.v. q24h for 4 days or vancomycin 1 g. q12h for up to 14 days.

The main criteria for evaluation will be:

* Efficacy
* Safety
* Microbiologic eradication

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained
2. Male or female ≥18 years of age
3. If female of childbearing potential, willing to practice reliable birth control measures and documented negative pregnancy test
4. Skin and skin structure infections of a complicated nature that require intravenous antibiotic treatment
5. Gram-positive infecting pathogen
6. Physician determination that vancomycin would be the initial treatment of choice
7. At least three clinical signs and symptoms associated with the cSSSI:

   * Pain;
   * Tenderness to palpation;
   * Elevated Temperature;
   * Elevated White blood count;
   * Swelling and/or induration;
   * Erythema (>1 cm beyond edge of wound or abscess);
   * Pus formation;
8. Creatinine clearance of ≥50 mL/min.

Exclusion Criteria:

1. MSSA
2. Known or suspected bacteremia, osteomyelitis, or endocarditis
3. Primary study infection of an uncomplicated nature such as furuncles, simple abscesses, cellulitis not requiring i.v., perirectal abscess, hidradenitis suppurativa, third degree burn infections or other minor infections;
4. Conditions where required surgery (in and of itself) constitutes curative treatment of the infection (e.g., amputation);
5. Necrotizing infections or concomitant gangrene;
6. Myositis with or without skin and skin structure infections;
7. Hemodialysis or peritoneal dialysis;
8. BMI ≥40 kg/m2;
9. Previous antibiotics exceeding 24 hours within the 48 hours prior to the first dose of study drug
10. Patients admitted for rhabdomyolysis including drug overdose
11. Neutropenic patients with absolute neutrophil count ≤500 cells/mm3
12. Known HIV-infected patients with CD4 count ≤200 cells/ mm3;
13. Baseline CPK values ≥2 X ULN (upper limit of normal);
14. Has received an investigational drug within 30 days of study entry;
15. Known to be allergic or intolerant to study medications;
16. unlikely to comply with study procedures
17. Is expected to receive HMG CoA Reductase Inhibitors from enrollment through End of Treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate at TOC

SECONDARY OUTCOMES:
difference between clinical response rates at EOT
microbiological eradication rates

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nathan, D.O., Principal Investigator — Idaho Falls Infectious Diseases, PLLC
Locations (1):
- Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho, United States

REFERENCES:
- [Derived] Katz DE, Lindfield KC, Steenbergen JN, Benziger DP, Blackerby KJ, Knapp AG, Martone WJ. A pilot study of high-dose short duration daptomycin for the treatment of patients with complicated skin and skin structure infections caused by gram-positive bacteria. Int J Clin Pract. 2008 Sep;62(9):1455-64. doi: 10.1111/j.1742-1241.2008.01854.x. Epub 2008 Jul 25. PMID 18662172